CLINICAL TRIAL: NCT01440010
Title: TARGeted Intraoperative radioTherapy With the INTRABEAM-System as an Advanced Boost in Patients With Breast Cancer - A Quality Control Registry in Germany (TARGIT BQR)
Brief Title: TARGeted Intraoperative radioTherapy With INTRABEAM as a Boost for Breast Cancer - A Quality Control Registry
Acronym: TARGIT_BQR
Status: Completed | Type: Observational
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Elena Sperk, MD, Senior Consultant, Managing Director Clinical Trials Unit Mannheim Cancer Center, Universitätsmedizin Mannheim
Other Study IDs: TARGIT BQR
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: IORT; Boost; Breast cancer; Local recurrence; Toxicity; LENT SOMA; TARGIT; Quality Control Registry
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IORT with 50 kV x-rays, 20 Gy: Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  Interventions: Radiation: IORT with 20 Gy

INTERVENTIONS:
Radiation: IORT with 20 Gy — Intraoperative radiotherapy with the INTRABEAM System with 20 Gy
  Other Names: Whole breast irradiation

SUMMARY:
Quality Control Registry for IORT used as an anticipiated boost with 20 Gy at the applicator surface followed by EBRT

DETAILED DESCRIPTION:
Quality Control Registry of a standard treatment with intraoperative radiotherapy during breast conserving surgery with 20 Gy at the applicator surface as an advanced boost followed by a shortened external beam radiotherapy. This is a prospective phase IV study to evaluate real life data of IORT Boost. Study runs in Germany with 13 active centers recruiting. Due to the nature of the study (registry) there is no need for randomization. Inclusion of n = >1000 patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* Tumor diameter < 3,5 cm
* Informed consent

Exclusion Criteria:

* No informed consent
* Tumor size > 3,5 cm
* No indication for a boost

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with breast cancer and a tumor diameter < 3,5 cm plannend for breast conserving surgery. Intraoperative radiotherapy (IORT) is applied as an advanced boost with 20 Gy at the applicator surface during surgery. Its feasibility was already shown. IORT as a boost is considered as one of several boost techniques in the S3-Leitlinie (national guideline) for breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1133 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sperk, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- University Medical Center Mannheim, Mannheim, Germany

REFERENCES:
- [Background] Andersen KG, Gartner R, Kroman N, Flyger H, Kehlet H. Persistent pain after targeted intraoperative radiotherapy (TARGIT) or external breast radiotherapy for breast cancer: a randomized trial. Breast. 2012 Feb;21(1):46-9. doi: 10.1016/j.breast.2011.07.011. Epub 2011 Aug 23. PMID 21865044
- [Background] Sautter-Bihl ML, Sedlmayer F, Budach W, Dunst J, Engenhart-Cabillic R, Fietkau R, Feyer P, Haase W, Harms W, Rodel C, Souchon R, Wenz F, Sauer R. Intraoperative radiotherapy as accelerated partial breast irradiation for early breast cancer : beware of one-stop shops? Strahlenther Onkol. 2010 Dec;186(12):651-7. doi: 10.1007/s00066-010-8001-2. PMID 21127826
- [Background] Vaidya JS, Baum M, Tobias JS, Wenz F, Massarut S, Keshtgar M, Hilaris B, Saunders C, Williams NR, Brew-Graves C, Corica T, Roncadin M, Kraus-Tiefenbacher U, Sutterlin M, Bulsara M, Joseph D. Long-term results of targeted intraoperative radiotherapy (Targit) boost during breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):1091-7. doi: 10.1016/j.ijrobp.2010.07.1996. Epub 2010 Oct 15. PMID 20951505
- [Background] Keshtgar MR, Vaidya JS, Tobias JS, Wenz F, Joseph D, Stacey C, Metaxas MG, Keller A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy for breast cancer in patients in whom external beam radiation is not possible. Int J Radiat Oncol Biol Phys. 2011 May 1;80(1):31-8. doi: 10.1016/j.ijrobp.2010.01.045. Epub 2010 Jun 18. PMID 20646864
- [Background] Vaidya JS, Joseph DJ, Tobias JS, Bulsara M, Wenz F, Saunders C, Alvarado M, Flyger HL, Massarut S, Eiermann W, Keshtgar M, Dewar J, Kraus-Tiefenbacher U, Sutterlin M, Esserman L, Holtveg HM, Roncadin M, Pigorsch S, Metaxas M, Falzon M, Matthews A, Corica T, Williams NR, Baum M. Targeted intraoperative radiotherapy versus whole breast radiotherapy for breast cancer (TARGIT-A trial): an international, prospective, randomised, non-inferiority phase 3 trial. Lancet. 2010 Jul 10;376(9735):91-102. doi: 10.1016/S0140-6736(10)60837-9. PMID 20570343
- [Background] Herskind C, Griebel J, Kraus-Tiefenbacher U, Wenz F. Sphere of equivalence--a novel target volume concept for intraoperative radiotherapy using low-energy X rays. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1575-81. doi: 10.1016/j.ijrobp.2008.08.009. PMID 19028280
- [Background] Belletti B, Vaidya JS, D'Andrea S, Entschladen F, Roncadin M, Lovat F, Berton S, Perin T, Candiani E, Reccanello S, Veronesi A, Canzonieri V, Trovo MG, Zaenker KS, Colombatti A, Baldassarre G, Massarut S. Targeted intraoperative radiotherapy impairs the stimulation of breast cancer cell proliferation and invasion caused by surgical wounding. Clin Cancer Res. 2008 Mar 1;14(5):1325-32. doi: 10.1158/1078-0432.CCR-07-4453. PMID 18316551
- [Background] Welzel G, Hofmann F, Blank E, Kraus-Tiefenbacher U, Hermann B, Sutterlin M, Wenz F. Health-related quality of life after breast-conserving surgery and intraoperative radiotherapy for breast cancer using low-kilovoltage X-rays. Ann Surg Oncol. 2010 Oct;17 Suppl 3:359-67. doi: 10.1245/s10434-010-1257-z. Epub 2010 Sep 19. PMID 20853059
- [Background] Kraus-Tiefenbacher U, Blank E, Wenz F. Intraoperative radiotherapy during a second breast-conserving procedure for relapsed breast cancer after previous external beam radiotherapy. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1279-80. doi: 10.1016/j.ijrobp.2011.02.038. No abstract available. PMID 21683889
- [Background] Wasser K, Ruch M, Brade J, Schoeber C, Kraus-Tiefenbacher U, Schnitzer A, Engel D, Wenz F, Sutterlin M, Schoenberg SO, Buesing KA. Do structural changes in the tumour bed after intraoperative radiotherapy (IORT) of breast cancer complicate the evaluation of mammograms in a long-term follow-up? Eur J Radiol. 2012 Mar;81(3):e255-9. doi: 10.1016/j.ejrad.2011.02.016. Epub 2011 Mar 4. PMID 21376493
- [Background] Blank E, Kraus-Tiefenbacher U, Welzel G, Keller A, Bohrer M, Sutterlin M, Wenz F. Single-center long-term follow-up after intraoperative radiotherapy as a boost during breast-conserving surgery using low-kilovoltage x-rays. Ann Surg Oncol. 2010 Oct;17 Suppl 3:352-8. doi: 10.1245/s10434-010-1265-z. Epub 2010 Sep 19. PMID 20853058
- [Background] Herskind C, Wenz F. Radiobiological comparison of hypofractionated accelerated partial-breast irradiation (APBI) and single-dose intraoperative radiotherapy (IORT) with 50-kV X-rays. Strahlenther Onkol. 2010 Aug;186(8):444-51. doi: 10.1007/s00066-010-2147-9. Epub 2010 Jul 29. PMID 20803285
- [Background] Wenz F, Welzel G, Blank E, Hermann B, Steil V, Sutterlin M, Kraus-Tiefenbacher U. Intraoperative radiotherapy as a boost during breast-conserving surgery using low-kilovoltage X-rays: the first 5 years of experience with a novel approach. Int J Radiat Oncol Biol Phys. 2010 Aug 1;77(5):1309-14. doi: 10.1016/j.ijrobp.2009.06.085. Epub 2010 Jan 25. PMID 20100643
- [Background] Ruch M, Brade J, Schoeber C, Kraus-Tiefenbacher U, Schnitzer A, Engel D, Wenz F, Sutterlin M, Schoenberg SO, Wasser K. Long-term follow-up-findings in mammography and ultrasound after intraoperative radiotherapy (IORT) for breast cancer. Breast. 2009 Oct;18(5):327-34. doi: 10.1016/j.breast.2009.09.010. PMID 19909898
- [Background] Kraus-Tiefenbacher U, Welzel G, Brade J, Hermann B, Siebenlist K, Wasser KS, Schneider FS, Sutterlin M, Wenz F. Postoperative seroma formation after intraoperative radiotherapy using low-kilovoltage X-rays given during breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2010 Jul 15;77(4):1140-5. doi: 10.1016/j.ijrobp.2009.06.008. Epub 2009 Oct 14. PMID 19836152
- [Background] Wenz F, Budach W, Dunst J, Feyer P, Haase W, Harms W, Sautter-Bihl ML, Sedlmayer F, Souchon R, Sauer R; DEGRO Expert Panel Breast Cancer. Accelerated partial-breast irradiation (APBI)--ready for prime time? Strahlenther Onkol. 2009 Oct;185(10):653-5. doi: 10.1007/s00066-009-8002-1. No abstract available. PMID 19806329
- [Background] Wenz F, Welzel G, Keller A, Blank E, Vorodi F, Herskind C, Tome O, Sutterlin M, Kraus-Tiefenbacher U. Early initiation of external beam radiotherapy (EBRT) may increase the risk of long-term toxicity in patients undergoing intraoperative radiotherapy (IORT) as a boost for breast cancer. Breast. 2008 Dec;17(6):617-22. doi: 10.1016/j.breast.2008.05.009. Epub 2008 Jul 22. PMID 18650091
- [Background] Kraus-Tiefenbacher U, Bauer L, Scheda A, Schoeber C, Schaefer J, Steil V, Wenz F. Intraoperative radiotherapy (IORT) is an option for patients with localized breast recurrences after previous external-beam radiotherapy. BMC Cancer. 2007 Sep 14;7:178. doi: 10.1186/1471-2407-7-178. PMID 17854511
- [Background] Wasser K, Schoeber C, Kraus-Tiefenbacher U, Bauer L, Brade J, Teubner J, Wenz F, Neff W. Early mammographic and sonographic findings after intraoperative radiotherapy (IORT) as a boost in patients with breast cancer. Eur Radiol. 2007 Jul;17(7):1865-74. doi: 10.1007/s00330-006-0556-z. Epub 2007 Jan 20. PMID 17237946
- [Background] Vaidya JS, Baum M, Tobias JS, Massarut S, Wenz F, Murphy O, Hilaris B, Houghton J, Saunders C, Corica T, Roncadin M, Kraus-Tiefenbacher U, Melchaert F, Keshtgar M, Sainsbury R, Douek M, Harrison E, Thompson A, Joseph D. Targeted intraoperative radiotherapy (TARGIT) yields very low recurrence rates when given as a boost. Int J Radiat Oncol Biol Phys. 2006 Dec 1;66(5):1335-8. doi: 10.1016/j.ijrobp.2006.07.1378. Epub 2006 Nov 2. PMID 17084562
- [Background] Kraus-Tiefenbacher U, Bauer L, Scheda A, Fleckenstein K, Keller A, Herskind C, Steil V, Melchert F, Wenz F. Long-term toxicity of an intraoperative radiotherapy boost using low energy X-rays during breast-conserving surgery. Int J Radiat Oncol Biol Phys. 2006 Oct 1;66(2):377-81. doi: 10.1016/j.ijrobp.2006.05.042. Epub 2006 Aug 2. PMID 16887294
- [Background] Kraus-Tiefenbacher U, Bauer L, Kehrer T, Hermann B, Melchert F, Wenz F. Intraoperative radiotherapy (IORT) as a boost in patients with early-stage breast cancer -- acute toxicity. Onkologie. 2006 Mar;29(3):77-82. doi: 10.1159/000091160. Epub 2006 Mar 3. PMID 16514267
- [Background] Kraus-Tiefenbacher U, Scheda A, Steil V, Hermann B, Kehrer T, Bauer L, Melchert F, Wenz F. Intraoperative radiotherapy (IORT) for breast cancer using the Intrabeam system. Tumori. 2005 Jul-Aug;91(4):339-45. doi: 10.1177/030089160509100411. PMID 16277101
- [Background] Pez M, Keller A, Welzel G, Abo-Madyan Y, Ehmann M, Tuschy B, Berlit S, Sutterlin M, Wenz F, Giordano FA, Sperk E. Long-term outcome after intraoperative radiotherapy as a boost in breast cancer. Strahlenther Onkol. 2020 Apr;196(4):349-355. doi: 10.1007/s00066-019-01525-7. Epub 2019 Oct 22. PMID 31641788
- [Derived] Goerdt L, Poemsl J, Spaich S, Welzel G, Abo-Madyan Y, Ehmann M, Berlit S, Tuschy B, Sutterlin M, Wenz F, Sperk E. Longitudinal cosmetic outcome after planned IORT boost with low kV X-rays-monocentric results from the TARGIT BQR registry. Transl Cancer Res. 2023 Jul 31;12(7):1715-1726. doi: 10.21037/tcr-23-88. Epub 2023 Jun 27. PMID 37588731

RESULTS

PARTICIPANT FLOW:
Groups:
- IORT With 50 kV X-rays, 20 Gy: Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  IORT with 50 kV x-rays, 20 Gy: Intraoperative radiotherapy with the INTRABEAM System with 20 Gy
Period: Overall Study
Arm/Group | IORT With 50 kV X-rays, 20 Gy
Started | 1133
Completed | 902
Not Completed | 231

BASELINE CHARACTERISTICS:
Population: 902 with complete paper work and minimum follow-up data set
Groups:
- IORT Boost With 20 Gy and Standard Whole Breast Irradition: All patients gave their informed consent prior to surgery and were planned for an anticipated boost immediately after tumor resection. Additionally, all patients were planned for standard whole breast radiotherapy with external beam radiation (EBRT). IORT with low-kV x-rays was given immediately after tumor resection into the tumorbed with 12-20 Gy as a single fraction with the INTRABEAM® system. EBRT was given according to standard of care procedures with conventional or hypofractioned schedules.
Arm/Group | IORT Boost With 20 Gy and Standard Whole Breast Irradition
Number analyzed (Participants) | 902
Age, Continuous [Median (Full Range); unit: years] | 61 [30 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 902
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Local Recurrence
Description: The follow-up was carried out every six months for the first two years, and then once a year. The follow-up always included a mammography in addition to a clinical examination. Kaplan-Meier-estimates were done to calculate the local recurrence rate
Time Frame: 5 years
Population: Planned IORT Boost plus whole breast irradiation
Measure: Number; unit: participants
Groups:
- IORT Boost: Planned IORT as Boost plus whole breast irradiation
Arm/Group | IORT Boost
Number analyzed (Participants) | 902
participants | 10

2. Secondary Outcome: Percentage of Patients With Chronic Higher Grade Fibrosis After IORT Boost
Description: Follow-up for toxicity assessment (LENT SOMA criteria: fibrosis, teleangiectasia, retraction, pain, breast edema, lymphedema, hyperpigmentation, ulceration) and oncological data took place before surgery, 6 weeks to 90 days after EBRT, 6 months after IORT, and then annually using standardized case report forms (CRFs).
Time Frame: 84 months
Population: Chronic higher grade fibrosis was defined as fibrosis grade 2 or higher occuring at least 3 times during follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | IORT Boost
Number analyzed (Participants) | 813
Participants | 132

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | IORT Boost With 20 Gy and Standard Whole Breast Irradition
All-Cause Mortality (participants affected / at risk) | 16/902
Serious Adverse Events (participants affected / at risk) | 0/902
Other Adverse Events (participants affected / at risk) | 83/902
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IORT Boost With 20 Gy and Standard Whole Breast Irradition (N=902)
Erythema (Skin and subcutaneous tissue disorders) | 40 (40) — Erythema
Palpable seroma (Skin and subcutaneous tissue disorders) | 83 (83) — Palpable seroma during follow-up.

LIMITATIONS AND CAVEATS:
902 patients were available for any analysis. Be aware that 8 patients with both sided cancers were included. So there were 910 affected breasts in 902 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-07-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT01440010/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT01440010/SAP_001.pdf